CLINICAL TRIAL: NCT03712202
Title: A Phase 2 Front-Line PET/CT-2 Response-Adapted Brentuximab Vedotin and Nivolumab Incorporated and Radiation-Free Management of Early Stage Classical Hodgkin Lymphoma (cHL)
Brief Title: Brentuximab Vedotin and Nivolumab in Treating Patients With Early Stage Classic Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18157; NCI-2018-01592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18157 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-08-06; First posted 2018-10-19 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Ann Arbor Stage I Hodgkin Lymphoma; Ann Arbor Stage I Mixed Cellularity Classic Hodgkin Lymphoma; Ann Arbor Stage I Nodular Sclerosis Classic Hodgkin Lymphoma; Ann Arbor Stage IA Hodgkin Lymphoma; Ann Arbor Stage IB Hodgkin Lymphoma; Ann Arbor Stage II Hodgkin Lymphoma; Ann Arbor Stage IIA Hodgkin Lymphoma; Ann Arbor Stage IIB Hodgkin Lymphoma; Classic Hodgkin Lymphoma; Lymphocyte-Rich Classic Hodgkin Lymphoma; Ann Arbor Stage I Lymphocyte-Depleted Classic HL; Ann Arbor Stage II Lymphocyte-Depleted Classic HL; Ann Arbor Stage II Mixed Cellularity Classic HL; Ann Arbor Stage II Nodular Sclerosis Classic HL
MeSH Terms: conditions — Hodgkin Disease | interventions — Bleomycin; Brentuximab Vedotin; Dacarbazine; Doxorubicin; Nivolumab; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I Arm A (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Biological: Nivolumab; Other: Quality-of-Life Assessment
- Group I Arm B (ABVD, nivolumab) (Experimental): Patients receive doxorubicin IV, bleomycin IV, vinblastine IV, dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 60 minutes on day 1. Treatment with nivolumab repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bleomycin; Drug: Dacarbazine; Drug: Doxorubicin; Biological: Nivolumab; Other: Quality-of-Life Assessment; Drug: Vinblastine
- Group II (AVD, brentuximab vedotin, nivolumab) (Experimental): Patients receive doxorubicin IV, vinblastine IV, dacarbazine, IV and brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients that are PET/CT negative receive nivolumab IV over 60 minutes on day 1. Treatment with nivolumab repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Dacarbazine; Drug: Doxorubicin; Biological: Nivolumab; Other: Quality-of-Life Assessment; Drug: Vinblastine

INTERVENTIONS:
Drug: Bleomycin — Given IV
  Other Names: BLEO; BLM
  Arms: Group I Arm B (ABVD, nivolumab)
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
  Arms: Group I Arm A (brentuximab vedotin, nivolumab); Group II (AVD, brentuximab vedotin, nivolumab)
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
  Arms: Group I Arm B (ABVD, nivolumab); Group II (AVD, brentuximab vedotin, nivolumab)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Group I Arm B (ABVD, nivolumab); Group II (AVD, brentuximab vedotin, nivolumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB
  Arms: Group I Arm B (ABVD, nivolumab); Group II (AVD, brentuximab vedotin, nivolumab)

SUMMARY:
This phase II trial studies how well brentuximab vedotin and nivolumab work in treating patients with stage I-II classic Hodgkin lymphoma. Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in a targeted way and delivers vedotin to kill them. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the 18-month progression free survival (PFS) for each arm of therapy stratified by positron emission tomography (PET)/computed tomography (CT)-2 response.

SECONDARY OBJECTIVES:

I. Assess safety, tolerability, and quality of life (QOL) for each arm of therapy.

II. Measure PET/CT-2 negativity rate after 2 lead-in cycles of standard of care doxorubicin, bleomycin, vinblastine, dacarbazine (ABVD).

III. Evaluate the 3-year PFS and overall survival (OS) for each arm of treatment.

EXPLORATORY OBJECTIVES:

I. Evaluate if a baseline antitumor immune response, as assessed by a Nanostring gene panel, correlates with PFS.

II. Evaluate if minimal residual disease (MRD) status, as monitored by cancer personalized profiling by deep sequencing (CAPP-Seq) of circulating tumor (ct) deoxyribonucleic acid (DNA), can be correlated with PFS.

OUTLINE: Patients are assigned to 1 of 2 groups based on their PET/CT-2 scans.

GROUP I (PET/CT-2 NEGATIVE): Patients without bulky disease are randomized to either Arm A or B and patients with bulky disease are assigned to Arm B.

ARM A: Patients receive brentuximab vedotin intravenously (IV) over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive doxorubicin IV, bleomycin IV, vinblastine IV, dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 60 minutes on day 1. Treatment with nivolumab repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

GROUP II (PET/CT-2 POSITIVE): Patients receive doxorubicin IV, vinblastine IV, dacarbazine, IV and brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients that are PET/CT negative receive nivolumab IV over 60 minutes on day 1. Treatment with nivolumab repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines.
* Eastern Cooperative Oncology Group (ECOG) =< 2.
* Histologically confirmed diagnosis of classical Hodgkin lymphoma (cHL) by current World Health Organization classification (nodular sclerosis, mixed cellularity, lymphocyte rich, lymphocyte depleted, or classical Hodgkin lymphoma, NOS [not otherwise specified]) at local enrolling center. Nodular lymphocyte-predominant Hodgkin lymphoma is excluded
* Stage IA, IB, IIA, or IIB cHL by Cotswold modified Ann Arbor staging done prior to any treatment with ABVD.
* Must have prior to standard of care ABVD treatment at least one lesion that is > 1.5 cm in the longest diameter on cross-sectional imaging and measureable in two perpendicular dimensions on CT and fludeoxyglucose (FDG) avid by PET.

Exclusion Criteria:

* Patients must be naive in terms of any prior therapy for Hodgkin lymphoma (including immunotherapy, chemotherapy or radiation therapy) with the exception that they may have received up to 2 cycles of ABVD as standard of care therapy prior to enrollment, as long as they can start protocol therapy (therapy administered in Arms A, B1/B2, or C) within timelines specified by the trial.
* Peripheral sensory neuropathy > grade 1 or any peripheral motor neuropathy.
* History of another primary malignancy that has not been in remission for at least 3 years. (The following are exempt from the 3-year limit: nonmelanoma skin cancer, fully excised melanoma in situ [Stage 0], curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolau [PAP] smear)
* Known cerebral/meningeal disease.
* History of progressive multifocal leukoencephalopathy (PML).
* Known history of pancreatitis.
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association class III-IV within 6 months prior to enrollment
* Uncontrolled cardiac disease including ventricular dysfunction, left ventricular ejection fraction < 45%, coronary artery disease, or arrhythmias.
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin, nivolumab, or any component of ABVD.
* Known active infection with hepatitis B or hepatitis C. Patients who are hepatitis B carriers can enroll if have a negative hepatitis B polymerase chain reaction (PCR) DNA test and are on hepatitis B suppressive medication management with entecavir or lamivudine. Patients with past active hepatitis C virus (HCV) infection are eligible if they are PCR negative after curative therapy. Testing to be done only in patients suspected of having infections or exposures.
* Known active infection with human immunodeficiency virus (HIV). Patients who are HIV positive can enroll if CD4 count is > 200/uL and have an undetectable or unquantifiable HIV viral load within 28 days of enrollment, have concurrent management with infectious disease specialists, and are on stable combination antiretroviral therapy. Participants are required to be on antiretroviral regimens that are in accordance with the current International acquired immune deficiency syndrome (AIDS) Society guidelines concurrently with chemotherapy. The specific agents are at the discretion of the Investigator and the use of investigational agents currently available on an expanded access basis is allowed. Use of experimental antiretroviral agents or those containing zidovudine (including Combivir and Trizivir) or ritonavir (includes Norvir or Kaletra), Cobicistat, Didanosine (Videx or Videx EC), or similar potent CYP3 inhibitors are prohibited. In order to be eligible, participants taking zidovudine or ritonavir, Cobicistat, Didanosine, or other CYP3 inhibitors must change to a different regimen 7 days prior to therapy initiation. Changes to highly active antiretroviral therapy (HAART) therapy during the study may be made if medically necessary (toxicity, failure of regimen, etc.). Participants must be on HAART for at least 7 days prior to therapy. HIV testing to be done only in patients suspected of having infections or exposures
* Subjects with active interstitial pneumonitis.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Females only: pregnant or breastfeeding.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
18-month Progression-free survival (PFS) for each arm of therapy | Up to 18 months
  Will be estimated using the method of Kaplan and Meier.

SECONDARY OUTCOMES:
Incidence of adverse events evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 | Up to 3 years
  Frequency tables will be used to summarize toxicity profile.
Scores from European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire C30, version 3 (EORTC-C30) for each arm of therapy | Up to 3 years
  All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Positron emission tomography/computed tomography-2 negativity rate | After 2 courses of ABVD (each course is 28 days)
  Will be estimated using the Deauville 5-point score/2014 Lugano Classsification
3-year PFS for each arm of treatment | Up to 3 years
  Will be estimated using the method of Kaplan and Meier.
Overall survival for each arm of treatment | Up to 3 years
  Will be estimated using the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (17):
- United States (17):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Medical Center, Duarte, California
  - University of California San Diego, San Diego, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYP/Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712